CLINICAL TRIAL: NCT03700112
Title: An Open Label, Randomized Crossover Study Comparing Nicotine Pharmacokinetics of Seven Electronic Cigarette Products and One Traditional Cigarette Across Two Delivery (10 Puff and Ad-libitum) Conditions, in Healthy Adult Smokers.
Brief Title: Clinical Study Comparing 7 ENDS Products and 1 Combustible Cigarette Using 2 Delivery Methods.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROT-00013
Record Dates: First submitted 2018-09-18; First posted 2018-10-09 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2019-01

CONDITIONS: Nicotine Dependence; Nicotine Dependence, Cigarettes; Tobacco Use; Tobacco Smoking
Keywords: Electronic Nicotine Delivery System; Combustible Cigarettes; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use; Tobacco Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- JUUL Virginia Tobacco flavored 5.0% ENDS (Experimental): Administration of JUUL Virginia Tobacco flavored 5.0% ENDS product consumed using 10 puffs delivery method
  Administration of JUUL Virginia Tobacco flavored 5.0% ENDS product consumed Ad-libitum delivery method
  Interventions: Other: JUUL Virginia Tobacco flavored 5.0% ENDS
- PMI iQOS Heat sticks (Experimental): Administration of PMI iQOS Heat sticks - Regular consumed using 10 puffs delivery method
  Administration of PMI iQOS Heat sticks - Regular consumed ad-libitum delivery method
  Interventions: Other: PMI iQOS Heat sticks
- Reynolds VUSE Solo ENDS - Original (Experimental): Administration of Reynolds VUSE Solo ENDS - Original consumed using 10 puffs delivery method
  Administration of Reynolds VUSE Solo ENDS - Original consumed using ad-libitum delivery method
  Interventions: Other: Reynolds VUSE Solo ENDS - Original
- Imperial MyBlu ENDS - Original (Experimental): Administration of Imperial MyBlu ENDS - Original consumed using 10 puffs delivery method
  Administration of Imperial MyBlu ENDS - Original consumed using ad-libitum delivery method
  Interventions: Other: Imperial MyBlu ENDS - Original
- Altria MarkTen ENDS - Bold Classic (Experimental): Administration of Altria MarkTen ENDS - Bold Classic consuming using 10 puffs delivery method
  Administration of Altria MarkTen ENDS - Bold Classic consuming using ad-libitum delivery method
  Interventions: Other: Altria MarkTen ENDS - Bold Classic
- MLV PHIX ENDS - Original Tobacco (Experimental): Administration of MLV PHIX ENDS - Original Tobacco consumed using 10 puffs delivery method
  Administration of with MLV PHIX ENDS - Original Tobacco consumed using ad-libitum delivery method
  Interventions: Other: MLV PHIX ENDS - Original Tobacco
- NJOY Daily EXTRA ENDS - Rich Tobacco (Experimental): Administration of NJOY Daily EXTRA ENDS - Rich Tobacco consumed using 10 puffs delivery method
  Administration of NJOY Daily EXTRA ENDS - Rich Tobacco consumed using delivery method and ad-libitum
  Interventions: Other: NJOY Daily EXTRA ENDS - Rich Tobacco
- Altria Marlboro combustible cigarette - Red (Experimental): Administration of Altria Marlboro combustible cigarette - Red consumed using 10 puffs delivery method Administration of Altria Marlboro combustible cigarette - Red consumed using ad-libitum delivery method
  Interventions: Other: Altria Marlboro combustible cigarette - Red

INTERVENTIONS:
Other: JUUL Virginia Tobacco flavored 5.0% ENDS — Virginia Tobacco Flavored 5.0% ENDS product is administered using a controlled method and adlibitum
  Arms: JUUL Virginia Tobacco flavored 5.0% ENDS
Other: PMI iQOS Heat sticks — PMI IQOS Heat sticks is administered using a controlled method and ad-libitum
  Arms: PMI iQOS Heat sticks
Other: Reynolds VUSE Solo ENDS - Original — Reynolds VUSE solo ENDS - Original is administered using a controlled method and ad-libitum
  Arms: Reynolds VUSE Solo ENDS - Original
Other: Imperial MyBlu ENDS - Original — Imperial MyBlu ENDS- original is administered using a controlled method and ad-libitum
  Arms: Imperial MyBlu ENDS - Original
Other: Altria MarkTen ENDS - Bold Classic — Altria MarkTen ENDS - Bold Classic is administered using a controlled method and ad-libitum
  Arms: Altria MarkTen ENDS - Bold Classic
Other: MLV PHIX ENDS - Original Tobacco — MLV PHIX ENDS - Original Tobacco is administered using a controlled method and ad-libitum
  Arms: MLV PHIX ENDS - Original Tobacco
Other: NJOY Daily EXTRA ENDS - Rich Tobacco — NJOY Daily EXTRA ENDS - Rich Tobacco is administered using a controlled method and ad-libitum
  Arms: NJOY Daily EXTRA ENDS - Rich Tobacco
Other: Altria Marlboro combustible cigarette - Red — Altria Marlboro combustible cigarette - Red is administered using a controlled method and ad-libitum
  Arms: Altria Marlboro combustible cigarette - Red

SUMMARY:
A Randomized Study Comparing Nicotine Pharmacokinetics of Seven Electronic Cigarette Products and One Traditional Cigarette Across Two Delivery (10 puff and ad- libitum) Conditions, in Healthy Adult Smokers

DETAILED DESCRIPTION:
E- cigarettes may be an acceptable alternative to traditional cigarette smoking. By utilizing vaporization rather than combustion, the generation and inhalation of HPHCs, smoke, and carbon monoxide (CO) may be reduced or avoided. This study will provide an understanding of the in vitro levels of nicotine obtained with use of the company's ENDS products compared to competitor products marketed in the United States of America (USA), and to a popular brand of combustible cigarette smoked in the USA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 60 years of age inclusive.
2. BMI between 18 to 35 kg / m2 inclusive.
3. Healthy based on medical history and screening assessments, in the opinion of the Investigator.
4. Current smoker of at least 8 cigarettes per day on average.
5. Has been smoking for at least 12 months prior to screening. Brief periods of non-smoking (e.g., up to ~7 consecutive days due to illness, trying to quit, participation in a study where smoking was prohibited) are permitted at the discretion of the Investigator.
6. Able to participate, and willing to give written informed consent and comply with study restrictions.

Exclusion Criteria:

1. Clinically relevant medical or psychiatric disorder, in the opinion of the Investigator.
2. Clinically significant abnormality on screening ECG.
3. Sustained blood pressure recordings at screening of < 90 mmHg or > 150 mmHg for systolic blood pressure, or < 50 mmHg or > 90 mmHg for diastolic blood pressure.
4. Sustained resting heart rate of > 100 or < 40 beats per minute at screening.
5. Positive result for urine drugs of abuse test or alcohol breath test at screening. If a positive urine drug test is observed, and it is believed the positive urine test is due to prescription drugs, the PI should obtain documentation that a) confirms the subject's use of the prescribed medication, and b) the prescribed medication will cause a false positive drug test.
6. Clinically significant abnormality in laboratory test results at screening, in the opinion of the Investigator.
7. Exposure to an investigational drug in a clinical trial within 1 month prior toAssessment Day 1.
8. Blood or plasma donation of > 500 mL within 1 month prior to Assessment Day 1.
9. Positive urine pregnancy test at screening or Assessment Day 1 in female subject.
10. Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-02-24 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Nicotine PK parameters will be calculated from the individual plasma concentrations per details provided in the SAP. | 48 days
  To estimate nicotine pharmacokinetics (PK) profiles across 8 E-Cigarette/cigarette products within-each and between-all delivery conditions (10 puffs versus ad libitum puffs) using Area Under the nicotine concentration-time curve (AUC1hour) calculated using linear trapezoidal summation from time zero (defined as the start of product use) to 60 minutes.
Nicotine PK parameters will be calculated from the individual plasma concentrations per details provided in the SAP. | 48 days
  Nicotine Pharmacokinetics (PK) profiles across 8 e-cigarettes/cigarette will be estimated using AUC1hour-baseline (baseline adjusted AUC1hour)
Nicotine PK parameters will be calculated from the individual plasma concentrations per details provided in the SAP. | 48 days
  Nicotine Pharmacokinetics (PK) profiles across 8 e-cigarettes/cigarette will be estimated using Cmax (Maximum measured plasma concentration over the duration of the measurement interval.
Nicotine PK parameters will be calculated from the individual plasma concentrations per details provided in the SAP. | 48 days
  Nicotine Pharmacokinetics (PK) profiles across 8 e-cigarettes/cigarette will be estimated using Cmax-baseline(Baseline adjusted Cmax)
Nicotine PK parameters will be calculated from the individual plasma concentrations per details provided in the SAP. | 48 days
  Nicotine Pharmacokinetics (PK) profiles across 8 e-cigarettes/cigarette will be estimated using Tmax(Time of the maximum measured plasma concentration over the duration of the measurement interval. If the maximum value occurs at more than one time point within the time span specified, Tmax is defined as the first time point with this value

SECONDARY OUTCOMES:
Measure exhaled Carbon Monoxide change in all product administration periods | 48 days
  To estimate change in exhaled carbon monoxide (CO) for 8 E-cigarettes/cigarettes Products, in all product administration periods under 2 different delivery (10 puff and ad-libitum) conditions. Exhaled CO will be measured 5-15 minutes prior to initiation of the first inhalation, and up to 15 minutes after the collection of the 30 minute PK sample
Characterize level of user Satisfaction for 8e-cigarette/cigarettes products using Modified Product Evaluation Scale | 48 days
  To characterize measures of subjective effects with use of 8 E-cigarettes/cigarettes Products under 2 different delivery (10 puff and ad-libitum) conditions using a modified Product Evaluations Scale questionnaire using scale below after collection of the 30-minute PK sample and exhaled CO measurement.
  Change in Evaluation: 1= not at all, 2= very little, 3= a little, 4= moderately, 5= a lot, 6= quite a lot, 7= extremely
  Four multi- item subscales will be derived from "Satisfaction" (questions 1, 2, 3, and 12); "Psychological Reward" (questions 4 through 8); "Aversion" (questions 9, 10, 16, and 18) and "Relief" (questions 11, 13, 14, 15, and reversed for question 19) and single questions 17 and 20 will be summarized.
Characterize consumption of 8 E-cigarettes/cigarettes products by collecting total number of puffs for each e-cigarette | 48 days
  To characterize consumptions of 8 E-cigarettes/cigarettes products within-each and between-all delivery conditions (10 puffs versus ad-libitum puffs), by collecting total number of puffs.

CONTACTS AND LOCATIONS:
Overall Officials: Concetta Carbonaro, Study Director — JUUL
Locations (1):
- Christchurch Clinical Studies Trust Ltd, Christchurch, New Zealand